CLINICAL TRIAL: NCT01306227
Title: L-Thyroxine Supplementation for Preterm Newborns Less Than 32 Weeks of Gestation With Transient Hypothyroxinemia of Prematurity: a Prospective Randomized Double-blind Trial
Brief Title: L-Thyroxine Supplementation for Preterm Newborns Less Than 32 Weeks of Gestation With Hypothyroxinemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRCIR07-DR-TOURNEUX
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Hypothyroxinemia
Keywords: Infant, newborn; Infant, preterm; Thyroid; Outcome; Newborns less than 32 weeks of gestation; TSH < 20 mIU/L and a FT4 < 0.80 ng/dL
MeSH Terms: conditions — Premature Birth; Thyroid Diseases | interventions — Thyroxine; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water (Placebo Comparator): Oral treatment with water for 6 weeks
  Interventions: Drug: water
- L-Thyroxine (Experimental): Oral treatment with L-Thyroxine for 6 weeks
  Interventions: Drug: L-Thyroxine

INTERVENTIONS:
Drug: L-Thyroxine — Treatment with L-Thyroxine:7,5 µg/kg/day. Oral treatment (one drop =5µg) in the morning, once a day.
  Arms: L-Thyroxine
Drug: water — Oral treatment with water. Equal number of drop of water as compared with the treatment arm (according to the body weight of the newborn) in the morning, once a day.
  Arms: water

SUMMARY:
Transient hypothyroxinemia of prematurity (THOP) is associated with neurodevelopmental impairment in preterm newborns < 32 weeks of gestation (WG). It is not known whether L-Thyroxine supplementation for preterm newborns <32 WG with THOP is beneficial.

The purpose of this study is to compare L-thyroxine treatment vs. placebo in newborn less than 32 WG with THOP.

The primary endpoint is the neurodevelopmental outcome at two years of life, assessed by the Brunet-Lézine score. The secondary endpoints are: death, bronchopulmonary dysplasia (oxygen therapy at 28 days of life and at 36 weeks of postnatal age), patent ductus arteriosus, shock requiring fluid loading or vasoactive treatments, enterocolitis, intraventricular hemorrhage, retinopathy of prematurity, deafness.

DETAILED DESCRIPTION:
Preterm newborns <32 weeks of gestation (WG) are screened for THOP between day 5 and day 7 of life. THOP is defined by thyroid-stimulating hormone (TSH) < 20 mIU/L and FT4 < 0.80 ng/dL. After obtaining written consent from the parents, preterm newborns <32 WG with THOP will be included. Randomization is stratified by center and 2 age-groups (24-28 WG and 29-32 WG). One arm will receive L-thyroxine treatment and the other arm will receive placebo. Treatment will be started within one week after diagnosis and will last 6 weeks. TSH and FT4 will be assayed 2 weeks after stopping treatment.

The primary endpoint is the neurodevelopmental outcome at two years of life, assessed by the Brunet-Lézine score.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 32 WG
* FT4 (5, 6 or 7 days of life) ≤ 0.8 ng/dL
* TSH (5, 6 or 7 days of life) < 20 mIU/L
* Written consent from the parents

Exclusion Criteria:

* Maternal thyroid disease
* FT4 (5, 6 or 7 days of life) > 0.8 ng/dL
* TSH (5, 6 or 7 days of life) > 20 mIU/L
* Grade III or IV intracerebral hemorrhage

Ages: 1 Week to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | 2 years old
  Brunet-Lézine score

SECONDARY OUTCOMES:
Morbidity associated with management of newborns < 32 WG with hypothyroxinemia | discharge, 1 year, 2 years
  * Death
  * Bronchopulmonary dysplasia (oxygen therapy at 28 days of life and at 36 weeks of postnatal age)
  * Patent ductus arteriosus,
  * Shock requiring fluid loading or vasoactive treatments
  * Enterocolitis
  * Intraventricular hemorrhage
  * Retinopathy of prematurity
  * Deafness

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tourneux, MD, Principal Investigator — Amiens University Hospital
Locations (3):
- France (3):
  - Caen University Hospital, Caen, Basse Normandie
  - Lens Hospital, Lens, Hauts-de-France
  - Amiens University Hospital, Amiens, Picardie